CLINICAL TRIAL: NCT02390817
Title: Effect of Sugammadex in Wakeup Procedure
Brief Title: Effect of Sugammadex for Muscle Motor Response and Awareness in Intraoperative Wakeup
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Collaborators: Private Ortopedia Hospital, Seyhan Adana (Other)
Responsible Party: Principal Investigator, ebru biricik, Anesthesiologist, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: wakeup01
Record Dates: First submitted 2015-02-12; First posted 2015-03-18 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2016-10

CONDITIONS: Spinal Curvatures
MeSH Terms: conditions — Spinal Curvatures | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Active Comparator): At the wakeup status Sugammadex 2 mg/kg single dose will perform.
  Interventions: Drug: Sugammadex
- Neostigmine (Placebo Comparator): At the wakeup status Neostigmine 0,04 mg/kg single dose will perform.
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Administration of Sugammadex
  Other Names: group I
  Arms: Sugammadex
Drug: Neostigmine — Administration of Neostigmine
  Other Names: group II
  Arms: Neostigmine

SUMMARY:
The study will be performed to evaluate motor response and awareness with using sugammadex during wakeup procedure in spine surgery. The investigator's goal is to investigate the effect of sugammadex on the state of consciousness and motor-somatosensorial evoked potentials.

DETAILED DESCRIPTION:
Between 10-25 age, American Society of Anesthesiologist clinical status(ASA) I-II, 60 patient which will be performed spine surgery in orthopedics clinic will be enrolled in this study. Patient will be randomized into two group that include 20 patient. General anesthesia will be administered by Totally intravenous anesthesia (TIVA) with propofol and remifentanyl for all patients. Two groups will be monitored with BIS (bispectral index), TOF (train-of-for) MEP (motor evoked potential) and SSEP (somatosensorial potential). During wakeup procedure, in group S, TIVA will be stopped and 2 mg/kg of sugammadex will be given intravenously. BIS, TOF, MEP, SSEP will be measured. In group N, TIVA will be stopped and 0.04 mg/kg of neostigmine will be given. Also BIS, TOF, MEP, SSEP will be measured. Sugammadex will be given group S and Neostigmine will be given group N at the end of the operation. At postoperative sixth hour, the investigators will visit all the patients and ask standard questions about intraoperative wakeup procedure.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) physical status I-II patients
* spine surgery
* 10-25 age

Exclusion Criteria:

* ASA III and above
* Patient refusal
* neuromuscular disease

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Time to consciousness | 30 min
  time to obeying verbal commands after reversal of NMBAs

SECONDARY OUTCOMES:
To assess Motor Evoked Potential values | 4 hours
  Motor Evoked Potential (MEP)
To assess Somatosensorial Evoked Potential values | 4 hours
  Somatosensorial Evoked Potential (SSEP)

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Biricik, Study Director — Medical Director
Locations (2):
- Turkey (Türkiye) (2):
  - Ebru Biricik, Adana, Sarıçam
  - Çukurova University, Adana, Çukurova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adamus M, Hrabalek L, Wanek T, Gabrhelik T, Zapletalova J. Intraoperative reversal of neuromuscular block with sugammadex or neostigmine during extreme lateral interbody fusion, a novel technique for spine surgery. J Anesth. 2011 Oct;25(5):716-20. doi: 10.1007/s00540-011-1209-1. Epub 2011 Aug 13. PMID 21842171
- See also: full text — http://pubmed.gov